CLINICAL TRIAL: NCT04224792
Title: Effects of Exercise Training on Fatigue in Thyroid Cancer Survivors
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to pandemic, unable to see patients
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, M. Regina Castro, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-008397
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Center-based exercise group (Experimental): Subjects will be enrolled into a center-based exercise program.
  Interventions: Other: Center-based exercise program
- Home-based exercise group (Experimental): Subjects will be enrolled into a home-based exercise program.
  Interventions: Other: Home-based exercise program

INTERVENTIONS:
Other: Center-based exercise program — A routine individualized exercise prescription and supervised exercise sessions at a minimum of once per week for 11 weeks with an exercise prescription updated monthly.
  Arms: Center-based exercise group
Other: Home-based exercise program — A one-time supervised exercise session with Cardiac Rehabilitation staff and a routine individualized exercise prescription for exercises to do at home. Additionally, weekly telephone followup calls by a clinical exercise physiologist for 11 weeks consisting of an exercise tip.
  Arms: Home-based exercise group

SUMMARY:
Researchers are trying to determine whether an exercise program reduces fatigue and improves physical activity in thyroid cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18yrs of age with well-differentiated thyroid cancer and self-reported fatigue any time after initial treatment of thyroid cancer.
* English speaking
* Able to provide consent

Exclusion Criteria:

* Pregnant
* Medullary thyroid cancer
* Anaplastic thyroid cancer
* Physical limitations to perform exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-30 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Fatigue symptoms | Baseline, 12 weeks
  Change in fatigue symptoms measured using the self-reported Fatigue Symptom Inventory (FSI) survey
Physical activity | Baseline, 12 weeks
  Change in physical activity measured using the self-reported International Physical Activity questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Regina Castro, MD, Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials